CLINICAL TRIAL: NCT03793387
Title: Preoperative Versus Intraoperative Transbronchial Dye Localization for Small Pulmonary Nodule : A Prospective Randomized Trial
Brief Title: Intra-op vs Pre-op Transbronchial Localization for Small Lung Nodule
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital Hsin-Chu Branch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 107-097-F
Record Dates: First submitted 2019-01-02; First posted 2019-01-04 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Pre-op (Experimental)
  Interventions: Procedure: AF-guided endobronchial marking
- Intra-op (Active Comparator)
  Interventions: Device: ENB-guided endobronchial marking

INTERVENTIONS:
Procedure: AF-guided endobronchial marking — Bronchoscopic dye marking under CBCT-augmented fluoroscopic guidance
  Arms: Pre-op
Device: ENB-guided endobronchial marking — Bronchoscopic dye marking with ENB system
  Arms: Intra-op

SUMMARY:
Comparing pre-operative transbronchial localization under augmented fluoroscopy and intra-operative transbronchial localization using electromagnetic navigation bronchoscopy system for small lung nodules.

DETAILED DESCRIPTION:
Using electromagnetic navigation bronchoscopy (ENB), transbronchial localization can be performed in the operating room (OR) under general anesthesia without extra radiation exposure, which is expected to reduce the discomfort for the patient during localization. This study will be carried out at the Hsinchu Branch of National Taiwan University Hospital. It is expected that 40 patients with pulmonary nodules will be randomly assigned into two groups. One group will receive bronchoscopic dye localization in the hybrid examination room equipped with cone-beam computed tomography, and the other group will receive ENB-guided dye localization in OR. The primary goal of the study was to compare the localization duration of the two groups of patients, the total dose of radiation exposure during localization and the incidence of location-related complications, and the secondary goals were the results of the surgical procedure, including the surgical duration.

ELIGIBILITY:
Inclusion Criteria:

A. One of each: lung nodule size less than 1 cm; depth more than 2 cm; GGO lesion B. 20~90 years old C. sign permit

Exclusion Criteria:

A. Previous emphysema, TB, COPD B. Previous ipsilateral thoracic surgery C. Bleeding tendency D. Heart failure, cirrhosis, CKD E. Pregnancy or breast feeding F. Immunocompromised G. Severe infection H. Unable to sign permit

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-07-08 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Successful localization | 2 days
  Discrepancy from lesion to marking: less than 1 cm
Successful resection | 2 days
  Lesion contained in first resected specimen

SECONDARY OUTCOMES:
Localization duration | 1 day
  Total time span of localization procedure
Total radiation exposure | 2 days
  Radiation during entire localization procedure
Complication | 14 days
  Procedure related complication

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Hsin-Chu Branch, Taipei, Hsin-Chu County, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided